CLINICAL TRIAL: NCT03067766
Title: A Pilot Study to Test the Feasibility of Comic Art Creation for Symptom Management in Cancer Supportive Care
Brief Title: Comic Art Creation as Supportive Care in Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16251; NCI-2017-00287 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16251 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Caregiver; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Art Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workshop A (10 weeks - comic art creation workshop) (Experimental): Patients and a family member, caretaker, or friend participate in an artist-led comic art therapy workshop over 2 hours once a week for 10 weeks. Patients and participants receive a range of assignments that focus on creative art and experimentation with materials and storytelling in order to make a series of small handmade books that relate directly or indirectly to their experience with cancer. Patients undergo a qualitative interview over approximately 45 minutes and complete validated questionnaires within 4 weeks prior to the workshop and midway through the workshop.
  Interventions: Procedure: Art Therapy; Other: Interview; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration
- Workshop B and C (5 weeks - comic art creation workshop) (Experimental): Patients participate in an artist-led comic art therapy workshop over 3 hours once a week for 5 weeks. Patients receive a range of assignments that focus on creative art and experimentation with materials and storytelling in order to make a series of small handmade books that relate directly or indirectly to their experience with cancer. Patients undergo a qualitative interview over approximately 45 minutes and complete validated questionnaires within 4 weeks prior to the workshop.
  Interventions: Procedure: Art Therapy; Other: Interview; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Art Therapy — Participate in a comic art creation workshop
Other: Interview — Undergo qualitative interviews
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well comic art creation works as supportive care in cancer patients and caregivers. Participating in a comic art creation workshop may help patients and their family members or friends share their medical experience through storytelling and drawings in a way that can, but does not have to, reflect the real world. It may also help improve emotional wellbeing and communication in cancer patients and caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of using a 10 week (Workshop A) or a 5 week (Workshops B-C) comic art creation workshops for supportive care.

II. To determine the feasibility of studying comic art creation workshops for supportive care.

III. To describe those factors affecting the ability or inability of participants to engage in the workshop.

SECONDARY OBJECTIVES:

I. To describe changes in emotional wellbeing and communication of patients and caretakers/family/friends.

TERTIARY OBJECTIVES:

I. Identify the methods that most engage supportive care patients and caretakers.

II. Identify the social and cultural interactions most impacted by comics creation.

III. To describe participant feedback regarding the intervention and study design.

OUTLINE: Patients are assigned to 1 of 2 arms.

WORKSHOP A: Patients and a family member, caretaker, or friend participate in an artist-led comic art therapy workshop over 2 hours once a week for 10 weeks. Patients and participants receive a range of assignments that focus on creative art and experimentation with materials and storytelling in order to make a series of small handmade books that relate directly or indirectly to their experience with cancer. Patients undergo a qualitative interview over approximately 45 minutes and complete validated questionnaires within 4 weeks prior to the workshop and midway through the workshop.

WORKSHOPS B AND C: Patients participate in an artist-led comic art therapy workshop over 3 hours once a week for 5 weeks. Patients receive a range of assignments that focus on creative art and experimentation with materials and storytelling in order to make a series of small handmade books that relate directly or indirectly to their experience with cancer. Patients undergo a qualitative interview over approximately 45 minutes and complete validated questionnaires within 4 weeks prior to the workshop.

After completion of the study, patients are followed up at 1 and 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant
* Workshop A (2017 - 10 weeks- City of Hope)

  * Either one of the following:
  * City of Hope (COH) cancer patient (all types and at any time point of their disease) OR
  * Caretaker/friend family member of the cancer patient
* Workshops B and C (2018 - 5 weeks - City of Hope)

  * Cancer patients (all types and at any time point in their disease)
  * Note: documentation to confirm this eligibility criteria will not be requested; self-reporting as a cancer patient will be considered adequate
* Ability read and speak English
* Willingness and ability to complete the entire workshop, including the interviews and questionnaires (there is no predetermined qualification with regard to the ability to hold an artist tool; accommodations and creative solutions will be made to facilitate participation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the comic art creation workshop defined as participant completion and psychosocial value of the comic art | Up to 1.5 years
  The project will be considered feasible if most of the participants complete the study and consider the comic art to have personal meaning, and if an initial power calculation indicates that a sufficiently powered randomized controlled trial is possible given the resources of the study team. It is anticipated that the psychosocial value of the art will be largely derived from the internal creation process and further assessment of the artistic products will not be conducted.

SECONDARY OUTCOMES:
Change in anxiety and depression as measured by the Hospital Anxiety and Depression Scale questionnaire | Baseline to up to 6 weeks post-workshop
  Statistical analysis will include Wilcoxon signed ranks test of pre, mid and post workshop HRQOL and symptom assessments. The Friedman test will be used to measure magnitude of difference within a case.
Change in health-related quality of life (HRQOL) as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 | Baseline to up to 6 weeks post-workshop
  Statistical analysis will include Wilcoxon signed ranks test of pre, mid and post workshop HRQOL and symptom assessments. The Friedman test will be used to measure magnitude of difference within a case.

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslava Salman, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States